CLINICAL TRIAL: NCT05839977
Title: Possibilities of Using Telerehabilitation for the Therapy of Balance and Walking Disorders in Patients With Multiple Sclerosis in Clinical Practice
Brief Title: The Effect of Telerehabilitation on Balance in People With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Barbora Staníčková, Possibilities of using telerehabilitation for the therapy of balance and walking disorders in patients with multiple sclerosis in clinical practice, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CharlesUniversity
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Telerehabilitation
Keywords: multiple sclerosis; telerehabilitation; remote rehabilitation; exergaming; balance
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individual telerehabilitation group (Experimental): 20 patients with multiple sclerosis
  Interventions: Other: Individual telerehabilitation
- Video based exercise group (Active Comparator): 20 patients with multiple sclerosis
  Interventions: Other: Home exercises based on videos
- Control group (No Intervention): 20 patients with multiple sclerosis

INTERVENTIONS:
Other: Individual telerehabilitation — The exercise will consist of strength and balance exercises using the Homebalance ® system
  Arms: Individual telerehabilitation group
Other: Home exercises based on videos — intervention include 12 video recordings of exercises created by a physiotherapist for home exercises, according to which they will also exercise
  Arms: Video based exercise group

SUMMARY:
The study will compare the effect of individual telerehabilitation with offline remote exercise through videos and with a control group without intervention. The monitored group will be people with multiple sclerosis with balance impairment. The duration of the intervention will be 12 weeks.

DETAILED DESCRIPTION:
Total of 60 persons will be randomly divided into two experimental and one control groups. After dividing into individual groups, all probands will be examined using objective and subjective tests for balance and walking. The same testing will be done after the end of the 12-week intervention.

The group with individual telerehabilitation will exercise twice a week. The exercise will consist of strength and balance exercises using the Homebalance ® system. For direct synchronous contact between the physiotherapist and the patient, an audiovisual link via the freely available ZOOM app was used.

The second experimental group will receive 12 video recordings of exercises created by a physiotherapist for home exercises, according to which they will also exercise twice a week.

The control group receives no intervention.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of definite MS
* subjectively perceived balance impairment
* clinically stable MS (at least 30 days since the last attack of the disease)
* ability to independently operate a PC or tablet, and

Exclusion Criteria:

* severe cognitive deficits that would interfere with understanding exercise instructions
* presence of other disease adversely affecting balance impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in balance (Berg Balance Scale) | Baseline to week 12
  Berg Balance Scale (BBS) is 14-item scale that evaluates balance.The 14 items are rated on either a 5-point (0-4) scale.
Change in functional mobility (Timed Up and Go) | Baseline to week 12
  Timed Up and Go test (TUG) is test used to measure functional mobility. The TUG test measures how long it takes to stand up, walk a distance of 3 metres, turn, walk back, and sit down again.
Change in functional mobility (Timed Up and Go Cognitive) | Baseline to week 12
  Timed Up and Go Cognitive (TUG Cognitive) is test used to measure functional mobility. The TUG test measures how long it takes to stand up, walk a distance of 3 metres, turn, walk back, and sit down again with an added cognitive task.
Change in balance (One leg stance) | Baseline to week 12
  One leg stance is test that evaluates balance. In the test, the time for which the tested person can stand on one leg is measured.

SECONDARY OUTCOMES:
Change in balance (Activity Balance Scale) | Baseline to week 12
  Activity Balance Scale (ABC Scale) is a patient-reported outcome measure that asks individuals to rate how confident they are that they will not lose their balance while performing 16 different activities.
Change in balance (Falls Efficacy Scale-I) | Baseline to week 12
  Falls Efficacy Scale-I (FES-I) is a questionnaire that assesses the fear of falling with a score ranging from minimum 16 (no concern about falling) to maximum 64 (severe concern about falling).
Change in walk (Multiple Sclerosis Walking Scale 12) | Baseline to week 12
  Multiple Sclerosis Walking Scale 12 (MSWS-12) is self-report measure of the impact of multiple sclerosis on the individuals walking ability. The questionnaire consists of 12 questions and scoring for each item is from 0 (no limitation) to 5 (extreme limitation).
Change in fatigue (Modified Fatigue Impact Scale) | Baseline to week 12
  Modified Fatigue Impact Scale (MFIS) is a questionnaire that assesses the impact of fatigue on physical, cognitive, and psychosocial functioning. MFIS consists of 21 items in scale 0-4 each item.

CONTACTS AND LOCATIONS:
Overall Officials: Barbora Staníčková, Mgr., Principal Investigator — First Faculty of Medicine, Charles University in Prague and General University Hospital
Locations (2):
- Czechia (2):
  - Center for Demyelinating Disease (RS Center), First Faculty of Medicine, Charles University and General University Hospital in Prague, Prague, Karlovo Náměstí 32
  - Department of Neurology and Center of Clinical Neuroscience, First Faculty of Medicine, Charles University and General University Hospital in Prague, Prague, Karlovo Náměstí 32